CLINICAL TRIAL: NCT05702710
Title: Percutaneous Internal Ring Suturing is a Safe and Effective Method in the Minimal Invasive Treatment of Inguinal Hernia in Neonates
Brief Title: Minimal Invasive Treatment of Inguinal Hernia in Neonates
Status: Completed | Type: Observational
Sponsor: Maltepe University (Other)
Responsible Party: Principal Investigator, Assoc. Prof. David T. Thomas, M.D., Associate Professor, Maltepe University
Other Study IDs: PIRS003
Record Dates: First submitted 2023-01-09; First posted 2023-01-27 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Inguinal Hernia; Surgery
MeSH Terms: conditions — Hernia, Inguinal | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Neonates Undergoing PIRS: All children <28 days of age undergoing PIRS for inguinal hernia repair
  Interventions: Other: Surgery (PIRS)

INTERVENTIONS:
Other: Surgery (PIRS) — Laparoscopic procedure for repair of inguinal hernia as described in:
  1) Thomas DT, Göcmen KB, Tulgar S, Boga I. Percutaneous internal ring suturing is a safe and effective method for the minimal invasive treatment of pediatric inguinal hernia: Experience with 250 cases. J Pediatr Surg. 2016 Aug;51(8):1330-5. doi: 10.1016/j.jpedsurg.2015.11.024. Epub 2015 Dec 11. PMID: 26777889.
  Other Names: Percutaneous Internal Ring Suturing

SUMMARY:
In this study, preoperative physical examination findings, peroperative findings and data, and postoperative follow-up results of newborns who underwent inguinal hernia repair with PIRS ("Percutaneous Internal Ring Suturing") method will be evaluated retrospectively.

DETAILED DESCRIPTION:
Congenital inguinal hernia is one of the most common surgical pathologies of childhood. Its treatment includes high ligation of the patent processus vaginalis by open or laparoscopic method. There are many described minimally invasive/laparoscopic repair techniques of inguinal hernias in children. One of them is "percutaneous internal ring suturing" or "Percutaneous Inner Ring Suturing".

There are many studies on the PIRS method in children. Two of these studies are prospective clinical studies published previously by the investigators of this study: in the first, the PIRS method was shown to be a safe and effective method for minimally invasive repair of inguinal hernia in children, and in the second, the use of subparalytic laryngeal masks in anesthesia of patients who underwent PIRS was shown to be sufficient for airway protection and anesthesia management in children undergoing laparoscopy.

Although there are many studies on the repair of inguinal hernia in children with PIRS or other minimally invasive methods in the last decade, there are very limited studies on the use of these methods in newborns, a special group of childhood patients. In the literature, there is no study examining only newborn patients. In this context, the study will be a first in the literature.

ELIGIBILITY:
Inclusion Criteria:

1. Having undergone PIRS surgery at the study institute between October 1, 2015 and January 1, 2023
2. Age between 0-28 days

Exclusion Criteria:

1. Age > 28 days
2. Having had surgery with open surgery
3. Having another surgical procedure performed in the same session

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Neonates <28 days of age undergoing PIRS
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2023-01-30 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
Surgery Time | Measured as time from skin prep until dressing is performed (approx. 20-30minutes)
  Time from skin prep to end of dressing
Anesthesia Time | Measured in minutes from induction to awakening (approx. 30-40minutes)
  Time from induction to awakening
Presence of Contralateral Patent Processus Vaginalis | Measured during surgery (approx. 5-10minutes)
  Whether a patent processus vaginalis was observed and repaired on laparoscopy

SECONDARY OUTCOMES:
Dose of Muscle Relaxant | Measured throughout surgery (20-30minutes)
  None, Subparalytic or Paralytic
Type of Airway Management Used | Measured throughout surgery (20-30minutes)
  ETT (Endotracheal Tube) or LMA (Laryngeal Mask Airway)

CONTACTS AND LOCATIONS:
Overall Officials: David T Thomas, MD, Principal Investigator — Maltepe University
Locations (1):
- Maltepe University Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Thomas DT, Gocmen KB, Tulgar S, Boga I. Percutaneous internal ring suturing is a safe and effective method for the minimal invasive treatment of pediatric inguinal hernia: Experience with 250 cases. J Pediatr Surg. 2016 Aug;51(8):1330-5. doi: 10.1016/j.jpedsurg.2015.11.024. Epub 2015 Dec 11. PMID 26777889
- [Background] Tulgar S, Boga I, Cakiroglu B, Thomas DT. Short-lasting pediatric laparoscopic surgery: Are muscle relaxants necessary? Endotracheal intubation vs. laryngeal mask airway. J Pediatr Surg. 2017 Nov;52(11):1705-1710. doi: 10.1016/j.jpedsurg.2017.02.010. Epub 2017 Feb 20. PMID 28249684
- [Background] Ergun E, Yagiz B, Kara YA, Abay AN, Balci O, Eryilmaz S, Ozguner IF, Karaman A, Karaman I. Comparison of laparoscopic percutaneous internal ring suturing method and open inguinal hernia repair in children under 3 months of age. Turk J Surg. 2021 Sep 28;37(3):215-221. doi: 10.47717/turkjsurg.2021.5157. eCollection 2021 Sep. PMID 35112055
- [Background] Wolak PK, Strzelecka A, Piotrowska-Gall A, Wolak PP, Piotrowska I, Dabrowska K, Wrobel J, Nowak-Starz G. Percutaneous Internal Ring Suturing (PIRS) - The Benefits of Laparoscopic Inguinal Hernia Repair. Ther Clin Risk Manag. 2022 Feb 22;18:135-144. doi: 10.2147/TCRM.S348197. eCollection 2022. PMID 35237037
- [Background] Pogorelic Z, Cohadzic T, Jukic M, Nevescanin Biliskov A. Percutaneous Internal Ring Suturing for the Minimal Invasive Treatment of Pediatric Inguinal Hernia: A 5-Year Single Surgeon Experience. Surg Laparosc Endosc Percutan Tech. 2021 Apr 15;31(2):150-154. doi: 10.1097/SLE.0000000000000878. PMID 33234851
- [Background] Wang F, Zhong H, Chen Y, Zhao J, Li Y, Chen J, Dong S. Single-site laparoscopic percutaneous extraperitoneal closure of the internal ring using an epidural and spinal needle: excellent results in 1464 children with inguinal hernia/hydrocele. Surg Endosc. 2017 Jul;31(7):2932-2938. doi: 10.1007/s00464-016-5309-8. Epub 2016 Nov 4. PMID 27815740